CLINICAL TRIAL: NCT05901818
Title: Safety and Efficacy of Autologous Induced Neural Stem Cell-derived Dopaminergic Precursor Cells in the Treatment of Parkinson's Disease
Brief Title: Safety and Efficacy of Autologous iNSC-DAP in the Treatment of Parkinson's Disease
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTC001
Record Dates: First submitted 2023-06-05; First posted 2023-06-13 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-05

CONDITIONS: Parkinson's Disease
Keywords: Autologous; iNSC; DA precursor cells; Parkinson's Disease; Cell therapy; Stereotaxic injection
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Autologous induced neural stem cell-derived DA precursor cells (Experimental): The patients will receive transplantation of autologous induced neural stem cell-derived DA precursor cells.
  Interventions: Drug: Autologous induced neural stem cell-derived DA precursor cells

INTERVENTIONS:
Drug: Autologous induced neural stem cell-derived DA precursor cells — The autologous induced neural stem cell-derived DA precursor cells will be stereotactically implanted into the striatum of PD patients.

SUMMARY:
This is a phase I, interventional, single arm, open-label, clinical study to evaluate the safety and efficacy of the striatal transplantation of autologous induced neural stem cell-derived DA precursor cells in Parkinson's Disease patients.

DETAILED DESCRIPTION:
Parkinson's Disease (PD) is the second most common neurodegenerative disease, caused by progressive depletion of midbrain dopaminergic neurons in the substantia nigra pars compacta. This clinical study will include the preparation of dopaminergic neural precursor cells derived from neural stem cells through reprogramming of patient's peripheral blood mononuclear cells (PBMCs), and transplantation of the obtained cells into the brains of PD patients by stereotaxic injection. Safety, tolerability, evidence of cell survival (using PET scan), and the efficacy on PD symptoms will be assessed at different time points up to 12 months post-transplantation.

ELIGIBILITY:
Inclusion Criteria:

Ages between 30 and 85 years, males or females; Diagnosed to be Parkinson's disease patients according to MDS Parkinson's disease diagnostic criteria; Disease history over 3 years; Hoehn and Yahr Stage less than or equal to 4 during the medication "on" time; Responsive to levodopa treatment (Maximum rate of improvement in MDS-UPDRS, part 3, is over 30%).

Exclusion Criteria:

Atypical Parkinsonian syndrome or secondary Parkinsonian syndrome; Accompanied with other central nervous system diseases; With other severe systemic diseases or dysfunction; With severe psychiatric disorders; Subjects are using hormone or cytotoxic drugs and cannot stop taking the drug during the trial; With cognitive disorders (MMSE<24); With severe dyskinesia (MDS-UPDRS part 4, score in 4.1/4.2 ≥ 2); Subjects have undergone previous brain surgery; Subjects are long-term user of anticoagulant; Subjects have intracranial lesions which may affect the surgery or follow-up studies as assessed by imaging; Subjects are unable to undergo MRI or AV133 PET examination; Pregnancy or in preparation for pregnancy; Not suitable to participate in this clinical trial as assessed by the study investigators/physicians.

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-06-13 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of changes during the medication "off" time in Movement Disorder Society-Sponsored Revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS), part III, in comparison with baseline values. | Within 12 months post-transplantation
  Minimum score: 0; Maximum score: 132; Higher scores mean a worse outcome.
Incidence and severity of transplant-related adverse events. | Within 12 months post-transplantation

SECONDARY OUTCOMES:
Assessment of changes in Movement Disorder Society-Sponsored Revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS), part I, in comparison with baseline values. | Within 12 months post-transplantation
  Minimum score: 0; Maximum score: 52; Higher scores mean a worse outcome.
Assessment of changes in Movement Disorder Society-Sponsored Revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS), part II, in comparison with baseline values. | Within 12 months post-transplantation
  Minimum score: 0; Maximum score: 52; Higher scores mean a worse outcome.
Assessment of changes in Movement Disorder Society-Sponsored Revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS), part IV, in comparison with baseline values. | Within 12 months post-transplantation
  Minimum score: 0; Maximum score: 24; Higher scores mean a worse outcome.
Assessment of changes during the medication "off" time in motor function by using Purdue Pegboard test and gait analyzer, in comparison with baseline values. | Within 12 months post-transplantation
Assessment of changes in the daily total medication "off" time in comparison with baseline values. | Within 12 months post-transplantation
Assessment of changes in Unified Dyskinesia Rating Scale in comparison with baseline values. | Within 12 months post-transplantation
  Minimum score: 0; Maximum score: 104; Higher scores mean a worse outcome.
Assessment of changes in daily levodopa-equivalent dose in comparison with baseline values. | Within 12 months post-transplantation
Assessment of changes in Parkinson's Disease Questionnaire (PDQ-39) in comparison with baseline values. | Within 12 months post-transplantation
Assessment of changes in AV133 PET imaging in comparison with baseline values. | Within 12 months post-transplantation
Assessment of changes in International Parkinson and Movement Disorder Society - Non-Motor Rating Scale (NMSS), in comparison with baseline values. | Within 12 months post-transplantation
  Minimum score: 0; Maximum score: 960; Higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital Capital Medical University, Beijing, Beijing Municipality, China